CLINICAL TRIAL: NCT00807079
Title: Phase I/II Study of Carboplatin in Association With Weekly Oral Topotecan in Patients With Metastatic or Recurrent Cervical Cancer
Brief Title: Carboplatin and Topotecan in Treating Patients With Relapsed or Metastatic Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000626790; ARCAGY-GINECO-CE102; ARCAGY-HYCAR; INCA-RECF0757; EUDRACT-2008-001842-19
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Carboplatin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: carboplatin; Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: carboplatin
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of topotecan when given together with carboplatin and to see how well they work in treating patients with relapsed or metastatic cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of topotecan hydrochloride when administered with carboplatin in patients with relapsed or metastatic cervical cancer. (Phase I)
* To determine the objective response rate in patients treated with this regimen. (Phase II)

Secondary

* To determine the dose-limiting toxicities of this regimen in these patients. (Phase I)
* To assess the progression-free survival of patients treated with this regimen. (Phase II)
* To assess the overall survival of patients treated with this regimen. (Phase II)
* To assess the tolerability of this regimen in these patients. (Phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study of topotecan hydrochloride followed by a phase II study.

Patients receive oral topotecan hydrochloride on days 1, 8, and 15 and carboplatin IV on day 1. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete a quality-of-life questionnaire at baseline and then every 3 months thereafter.

After completion of study therapy, patients are followed every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cervical cancer, including the following cell types:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Adenosquamous cell carcinoma
* Metastatic disease or in first relapse

  * Not curable by surgery and/or radiotherapy with or without chemotherapy
* At least 1 non-irradiated measurable lesion
* No CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Transaminases ≤ 3 times upper limit of normal (ULN) (≤ 5 times ULN in the presence of liver metastases)
* Total bilirubin ≤ 1.5 times ULN
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other cancer within the past 5 years except for adequately treated basal cell or squamous cell carcinoma of the skin
* No swallowing disorders or gastrointestinal disease resulting in an inability to take oral medication or a requirement for IV alimentation
* No altered intestinal absorption
* No peptic ulcers
* No nephrostomy

  * Double-J catheter allowed
* None of the following cardiovascular conditions within the past 6 months:

  * Uncontrolled hypertension
  * Coronary artery disease
  * NYHA class III or IV congestive heart failure
  * Ventricular arrhythmia
  * Unstable angina
  * Myocardial infarction
* No infection or serious illness that would preclude study treatment
* No contraindications to study treatment
* No psychological, familial, sociological, or geographical condition that would preclude follow-up

PRIOR CONCURRENT THERAPY:

* No prior cytotoxic therapy except for chemoradiotherapy or pelvic radiotherapy
* At least 6 months since prior platinum-based chemoradiotherapy
* No concurrent participation in another clinical trial that could interfere with the objectives of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of topotecan hydrochloride (Phase I) | 3 months
Objective response rate (Phase II) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Laure Chauvenet, MD, Principal Investigator — Hotel Dieu de Paris
Locations (1):
- Hotel Dieu de Paris, Paris, France